CLINICAL TRIAL: NCT05228769
Title: Evaluation of the Quality of Life After a Multidisciplinary Auditory Rehabilitation Program
Acronym: EQUAPRAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Sainte-Marie Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: EQUAPRAP
Record Dates: First submitted 2021-12-31; First posted 2022-02-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Acquired Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2008, the Handicap-Santé survey counted 10 million people with hearing difficulties in France, i.e. 16% of the national population. For 5.4 million of these people, the hearing limitations considered to be moderate to total, are likely to have repercussions on their daily life.

In 2010, 600,000 people with hearing loss wore hearing aids, including 360,000 with very severe to total limitations who were unable to follow a conversation with others.

Hearing loss can impact hearing skills (comprehension in noisy environments or with multiple speakers) and be a source of cognitive decline. It can also limit the quality of exchanges, communication and information taking.

Several studies have shown that hearing loss can also have a negative effect on quality of life, psychological well-being, personal fulfillment, social relationships and can lead to social isolation, depression and/or anxiety.

Currently, the treatment of people with hearing loss is often limited to hearing aids from a hearing aid specialist. Hearing rehabilitation and lip-reading training with a speech therapist may be offered at a later stage. However, many people who have been fitted with a hearing aid describe a decrease in their quality of life despite the fitting.

Current treatment seems to deal mainly with auditory-cognitive problems. To date, no multidisciplinary rehabilitation services seem to be offered in France to take into account the other consequences of this condition: anxiety, depression, and limitations in social participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age ≥ 18 years
* Patients with acquired hearing loss (mild, moderate, severe or profound)
* Patients with hearing aids
* Patients participating in a complete rehabilitation program
* Patients who master the French language

Exclusion Criteria:

* Patients with proven cognitive impairment
* Implanted patients
* Patients under guardianship or curatorship
* Patients deprived of liberty
* Patients under court protection
* Interruption of the rehabilitation program before a minimum of 6 half-days of HDJ
* Patients objecting to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired hearing loss (mild, moderate, severe or profound), with hearing aid, participating in a complete rehabilitation program between November 2015 and June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Impact of multidisciplinary rehabilitation on the quality of life of adults with hearing aids | Month 1
  This outcome corresponds to the Change in quality of life measured with the ERSA scale before and after rehabilitation.

SECONDARY OUTCOMES:
Patient profile of age | Month 1
  This outcome corresponds to the number of age categories
Patient profile of type of hearing loss | Month 1
  This outcome corresponds to the number of type of hearing loss.
Patient profile of severity | Month 1
  This outcome corresponds to the type of severity.
Quality of life of patients | Month 1
  This outcome corresponds to the overall quality of life, personal life, social life and work life of the assessment of the impact of deafness in adults. is a self-administered questionnaire. It is divided into 4 domains, each comprising 5 questions graded from 1 to 10. The questions are simple, and formulated so patients will answer according to how they feel at the actual time of the session.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SAFAR, MD, Principal Investigator — Hôpital Sainte-Marie
Locations (1):
- Hôpital Sainte-Marie, Paris, France

REFERENCES:
- [Background] Ciorba A, Bianchini C, Pelucchi S, Pastore A. The impact of hearing loss on the quality of life of elderly adults. Clin Interv Aging. 2012;7:159-63. doi: 10.2147/CIA.S26059. Epub 2012 Jun 15. PMID 22791988
- [Background] Brodie A, Smith B, Ray J. The impact of rehabilitation on quality of life after hearing loss: a systematic review. Eur Arch Otorhinolaryngol. 2018 Oct;275(10):2435-2440. doi: 10.1007/s00405-018-5100-7. Epub 2018 Aug 23. PMID 30159730